CLINICAL TRIAL: NCT07044648
Title: Middle Meningeal Artery Embolization for Treatment of Chronic Migraine: A Pilot Study
Brief Title: Middle Meningeal Artery Embolization for Chronic Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB submission never completed, study application withdrawn by IRB due to lack of response from PI
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00131621
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: chronic migraine; drug-resistant migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Middle Meningeal Artery Embolization (Experimental): Participants receive middle meningeal artery embolization
  Interventions: Procedure: Middle Meningeal Artery Embolization

INTERVENTIONS:
Procedure: Middle Meningeal Artery Embolization — Middle meningeal artery embolization using particles or coils

SUMMARY:
The main goal of this study is to find out how well middle meningeal artery coil embolization works for patients with recurrent chronic migraines that are not resolved with medication.

DETAILED DESCRIPTION:
This study seeks to evaluate the therapeutic potential of middle meningeal artery coil embolization as an interventional strategy for patients with recurrent and pharmacoresistant chronic migraine. Middle meningeal artery embolization has recently gained recognition as a safe and effective intervention for the management of chronic subdural hematoma, demonstrating a low complication profile. The procedure achieves therapeutic effect by reducing or occluding arterial flow within the middle meningeal artery, thereby minimizing arterial dilatation and facilitating hematoma resorption over time.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of migraine with or without aura, chronic migraine, unilateral or bilateral, moderate to severe intensity, 4-72 hours, familiar or sporadic, status migrainosus, primary or secondary
* Patient who failed pharmacologic treatment (at least 2 failed drugs treatment for more than 3 months) or have considerable side effects
* Patient with diagnosis of migraine and preference for embolization treatment
* Clinical follow up of at least 3 months
* Baseline computed tomography head (CTH) or MR brain which rule out additional intracranial pathology (patient with baseline intracranial pathology other than migraine will be excluded; see the exclusion criteria section below)
* Presence of patent middle meningeal artery homolateral to the side of migraine

Exclusion Criteria:

* Previous middle meningeal artery embolization for subdural hematoma
* Previous craniotomy
* Patients aged 17 years or younger.
* Incomplete embolization of middle meningeal artery
* Patient with baseline CTH or MR brain showing baseline intracranial pathology that can explain migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Migraine Disability Assessment (MIDAS) | Baseline
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Disability Assessment (MIDAS) | 1 Hour Post Procedure
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Disability Assessment (MIDAS) | Day 15 Follow Up
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Disability Assessment (MIDAS) | Month 3 Follow Up
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Disability Assessment (MIDAS) | Month 6 Follow Up
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Disability Assessment (MIDAS) | Month 12 Follow Up
  The MIDAS is a 7 item survey. Score range is Grade I-IV with a higher score indicating severe disabling headache.
Migraine Pain Scale | Baseline
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.
Migraine Pain Scale | 1 Hour Post Procedure
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.
Migraine Pain Scale | Day 15 Follow Up
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.
Migraine Pain Scale | Month 3 Follow Up
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.
Migraine Pain Scale | Month 6 Follow Up
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.
Migraine Pain Scale | Month 12 Follow Up
  Migraine pain scale range is 1-10 with a higher indicating severe level of pain.

SECONDARY OUTCOMES:
Number of Pain Meds Used Post Procedure | 1 Hour Post Procedure
  Number of pain meds used by participant post embolization procedure
Number of Pain Meds Used Post Procedure | 6 Hours Post Procedure
  Number of pain meds used by participant post embolization procedure
Number of Pain Meds Used Post Procedure | Day 15 Follow Up
  Number of migraine pain meds used by participant post embolization procedure
Number of Pain Meds Used Post Procedure | Month 3 Follow Up
  Number of migraine pain meds used by participant post embolization procedure
Number of Pain Meds Used Post Procedure | Month 6 Follow Up
  Number of migraine pain meds used by participant post embolization procedure
Number of Pain Meds Used Post Procedure | Month 12 Follow Up
  Number of migraine pain meds used by participant post embolization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hamad Farhat, MD, Principal Investigator — advocate christ medical center

IPD SHARING:
Plan to Share IPD: No